CLINICAL TRIAL: NCT00283894
Title: The Role of the Orexin System in Body Weight Regulation: Patients With Narcolepsy
Brief Title: Body Weight Regulation in Patients With Narcolepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060079; 06-DK-0079
Record Dates: First submitted 2006-01-29; First posted 2006-01-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-06-19

CONDITIONS: Narcolepsy
Keywords: Obesity; Leptin; Sleep Attacks; Energy Metabolism; Healthy Control; Narcolepsy; Healthy Volunteer; HV
MeSH Terms: conditions — Narcolepsy; Obesity

SUMMARY:
This study will measure energy expenditure (the rate at which the body burns calories), physical activity and caloric intake in people with narcolepsy to learn more about how the risk of becoming overweight or diabetic may be affected.

Healthy control subjects and people with narcolepsy between 18 and 55 years of age may be eligible for this study. Participants are withdrawn from their narcolepsy medication and undergo the following tests and procedures over 5 weeks before resuming medications.

* Blood draw for genetic studies.
* Collection of a cerebrospinal fluid sample.
* Diet to keep subjects' weight constant.
* Activity watch, using a device worn on the wrist to measure amount of movement, and an activity monitor worn at the waist to measure physical activity and caloric expenditure.
* Questionnaires about sleepiness, symptoms, food intake, exercise and mood.
* 24-hour urine collection and 24-hour blood draw to measure hormones.
* Glucose tolerance test. The subject drinks a sugar solution and blood samples are collected through a catheter before drinking the solution and 30 minutes, 1, 2 and 3 hours after drinking it.
* Startle reflex test. Subjects hear a loud noise through headphones and are asked to look at pictures.
* Sleep study to evaluate sleep-related breathing disturbances and record information about sleep stages.
* Indirect calorimetry test to measure how fast the body uses calories. A plastic canopy is placed over the face for several minutes to capture the air exhaled to analyze oxygen use. To measure the energy associated with meals, the same measurements are taken after the subject eats lunch.
* CT scan of the abdomen to see how much fat is deposited in the abdomen, and DEXA scan of the whole body to see the percentage of fat and muscle.
* Plethysmography. Participants sit in an enclosed chamber while the mass and volume of the body are measured by changes in air pressure.
* Neuropsychological testing to assess thought processes.
* Continuous 24-hour heart rate measurement.
* Metabolic chamber. Subjects spend 24 hours in a small room to measure the amount of oxygen inhaled and carbon dioxide exhaled.
* Walking/running test to assess level of physical conditioning.
* Dexamethasone CRH (corticotropin-releasing hormone) suppression test and CRH stimulation test. Subjects receive eight doses of 0.5 mg dexamethasone every 6 hours for a day and a half. After the last dose, two blood samples are drawn, then a dose of CRH is injected, and then six more blood samples are drawn over the next 3 hours.
* TRH (thyrotropin-releasing hormone) stimulation test. Subjects are given TRH through a vein, and several blood samples are then drawn over the next 3 hours.
* Doubly labeled water test. Subjects drink a dose of "heavy" water. Urine samples are collected at 2, 3 and 5 hours after drinking and again for two 4-hour collections a week later.

DETAILED DESCRIPTION:
BACKGROUND: Several cross-sectional studies have suggested that subjects with narcolepsy have increased body mass index (BMI) and insulin resistance. These subjects exhibit a decrease in cerebrospinal fluid (CSF) orexin levels, which has been causally linked to the clinical manifestations of this disease. Orexins are peptides expressed in a brain region, the lateral hypothalamic area, which stimulate appetite and modulate sleep. Low CSF orexin levels provoke narcolepsy-like behavior, such as excessive daytime sleepiness and a sudden loss of muscle tone known as cataplexy.

OBJECTIVES: The primary objective of this study is to determine whether subjects with narcolepsy have lower energy expenditure compared to healthy matched controls. In addition, we will assess food intake, physical activity, and other relevant parameters.

STUDY POPULATION: 18 to 55 year old men and premenopausal women with narcolepsy and healthy matched controls

DESIGN: This is a cross-sectional, case-controlled study of subjects with narcolepsy matched on a one-to-one basis with healthy, non-narcoleptic control subjects.

OUTCOME PARAMETERS: We will assess metabolic, hormonal, and energy expenditure parameters in subjects with narcolepsy. Outcomes: energy expenditure by various methods (indirect calorimetry, metabolic chamber, doubly-labeled water method); leptin circadian levels (frequent 24h sampling); physical activity, characterization of the main endocrine axes, and other relevant parameters.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients

-18 to 55 year old men and pre-menopausal women with current narcolepsy, otherwise healthy.

Controls

-18 to 55 year old healthy men and pre-menopausal women.

SUBJECTS WITH NARCOLEPSY INCLUSION:

* Having a current diagnosis of narcolepsy with moderate or severe daytime sleepiness for at least 6 months, according to the International Classification of Sleep Disorder (ICSD).
* Both new and previously diagnosed patients are eligible.
* Females of childbearing potential must have a negative serum pregnancy test.
* A valid barrier contraception method is required over the duration of the study.
* Patients must agree to refrain from operating a motor vehicle and from being involved in any other potentially hazardous activity during the tapering off and the drug-free periods.

SUBJECTS WITH NARCOLEPSY EXCLUSION:

* Pregnancy and lactation (women only)
* Use of birth control pills
* Menopause, defined as 6 consecutive months without mensis
* Clinical diagnosis of polycystic ovary disease, chronic history of anovulatory cycles or other alterations of the menstrual cycle (for women only)
* Use of any experimental drug or current participation in another research protocol
* Chronic amphetamines in the last 2 months and any drug known to influence the autonomic nervous system including appetite suppressants
* Excessive daytime sleepiness (EDS) related to:
* Sleep apnea
* Periodic limb movements
* Substance disorder or alcohol consumption
* Any concurrent psychiatric, neurological, neoplastic, endocrinologic, or infectious disease that may contribute to EDS
* Insufficient sleep (less than 6 hours/night) or any other known cause inducing sleepiness
* Working in an occupational environment that requires variable or routine night shifts
* History of head trauma or history of seizure
* Agitated state or severe anxiety, moderate or severe psychosis or dementia
* Current major depression (Hamilton score greater than 18), subjects currently receiving pharmacological treatment for depression (even if their Hamilton score is lower than 18), anyone who has or had suicidal ideation
* Dyskinesia or other neurological conditions
* Use of any medications that may influence sleep or contribute to EDS, except for anticataplectic medications, including:

Hypnotic, anxiolytic, chronic amphetamine use, antidepressants, antihistamine, clonidine, anticonvulsants

* Hyperthyroidism or hypothyroidism
* Symptomatic cardiac disease
* For those subjects consenting to the exercise test (Cooper test)

Any medical contraindication to exercise of moderate intensity and short duration including cardiovascular or respiratory conditions, morbid obesity, and severe osteoarthritis of the lower extremities

* Chronic illicit drug use
* Use of antipsychotic drugs
* Narcoleptic subjects with coexistent significant sleep apnea or respiratory disturbances are excluded
* Major cardiac rhythm disturbances, respiratory rate alterations, or any other major organ disease that would make the interpretation of HRV data arduous
* Fever

EXCLUSION RELATED TO THE METABOLIC STATUS:

* Weight fluctuations defined as increase or decrease in body weight greater than 5% over the last 3 months
* Unstable physical activity in the 3 months prior to study entry
* Any secondary cause of obesity, including:
* Cushing syndrome, hypothyroidism, GH and testosterone deficiency, polycystic ovarian syndrome, insulinoma, hypothalamic lesions, and genetic obesity syndromes such as Prader-Willy and other genetic syndromes
* Obesity-related medical conditions requiring pharmacological treatment
* Insulin-dependent diabetes mellitus
* Uncontrolled hypertension
* Uncontrolled hyperlipidemia
* Current smoking, defined as more than 2 cigarettes/day
* Strict vegetarian diet, defined as lack of milk, eggs, and diary products

HEALTHY CONTROL SUBJECT INCLUSION/EXCLUSION:

-In addition to the criteria specified above, healthy controls must be in good physical health and not on chronic medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01-20; Study Completion 2013-06-19

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cizza, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Blanco M, Gallego R, Garcia-Caballero T, Dieguez C, Beiras A. Cellular localization of orexins in human anterior pituitary. Histochem Cell Biol. 2003 Oct;120(4):259-64. doi: 10.1007/s00418-003-0562-z. Epub 2003 Aug 28. PMID 14574580
- [Background] Buchholz K, Schachinger H, Wagner M, Schorr U, Sharma AM, Deter HC. Enhanced affective startle modulation in salt-sensitive subjects. Hypertension. 2001 Dec 1;38(6):1325-9. doi: 10.1161/hy1101.096055. PMID 11751712
- [Background] Chabas D, Taheri S, Renier C, Mignot E. The genetics of narcolepsy. Annu Rev Genomics Hum Genet. 2003;4:459-83. doi: 10.1146/annurev.genom.4.070802.110432. PMID 14527309